CLINICAL TRIAL: NCT01528098
Title: Efficacy of Bisacodyl Given as Part of a Polyethylene Glycol-based Bowel Preparation Prior to Colonoscopy in Hospitalized Patients
Brief Title: Comparison of Bowel Cleansing Methods for Colonoscopy in Hospitalized Patients
Acronym: PEG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kangbuk Samsung Hospital (Other)
Collaborators: Soon Chun Hyang University (Other); Kyunghee University (Other); Hanyang University (Other)
Responsible Party: Principal Investigator, Dong Il Park, M.D, Ph.D., Associate professor, Department of Internal Medicine, Kangbuk Samsung Hospital
Other Study IDs: PEGPD
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Intestine; Complaints
Keywords: polyethylene glycol; bisacodyl

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PEG plus bisacodyl: Those who taken PEG 4L + bisacodyl 10mg
- PEG 4L: Those who taken PEG 4L alone

SUMMARY:
The purpose of this study is to compare two regimens of polyethylene glycol(PEG) plus bisacodyl versus PEG alone for bowel preparation in hospitalized patients.

DETAILED DESCRIPTION:
Inadequate bowel preparation may lead to a longer colonoscopy, and to an inability to identify lesions. PEG can provide a rapid orthograde peroral approach to colonic lavage without producing significant fluid or electrolyte changes. Thus PEG is now commonly used for bowel preparation. However, large amounts and unsatisfactory taste of PEG solution are generally poorly tolerated, especially in hospitalized patients who had comorbidity and restricted ambulation. Recently, a new PEG-based bowel cleansing agents became available. It combines PEG with a high dose of ascorbic acid or bisacodyl. Although many studies reported the efficacy of these combined solution for colonoscopy, but efficacy in hospitalized patients was under-recognized.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients for colonoscopy

Exclusion Criteria:

* age under 20 years or over 80 years
* major psychiatric illness
* known allergy to PEG
* serious condition- severe cardiac, renal, or metabolic diseases
* partial colon resection
* current acute exacerbation of chronic inflammatory bowel disease
* functional constipation defined by Rome III diagnostic criteria

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients for colonoscopy in university hospital.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-07 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
The efficacy of bowel preparation | one day (after colonoscopy)
  Ottawa scale

SECONDARY OUTCOMES:
Patient's compliance and acceptability | one day (after injestion of preparation solution)
  acceptability, Visual Analogue Scale
Patient's compliance and acceptability (2) | one day (after injestion of preparation solution)
  stress for ingestion, Stress 0(not) - 4(severe)
Patient's compliance and acceptability (3) | one day (after colonoscopy)
  willingness for re-evaluation, 0(very willing) - 4(some)

CONTACTS AND LOCATIONS:
Overall Officials: Dong Il Park, Professor, Principal Investigator — Kangbuk Samsung Hospital